CLINICAL TRIAL: NCT06948201
Title: Inorganic Nitrate as a Treatment for ANOCA: NO-ANOCA
Acronym: NO-ANOCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Patricia Rodriguez Lozano, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 302494
Record Dates: First submitted 2025-04-16; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Coronary Microvascular Dysfunction (CMD); Angina Patients With Non-obstructive Coronary Artery Disease
Keywords: angina; ANOCA; Non-obstructive Coronary Artery Disease; CMD; Non-Obstructive CAD; Chest Pain in Women
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: single-site, double-blind, randomized crossover pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice followed by placebo (Other): 70mL Nitrate Rich Beetroot Juice for 14 days followed by placebo (70mL nitrate depleted beetroot juice) for 14 days
  Interventions: Dietary Supplement: 70mL Nitrate Rich Beetroot Juice followed by placebo (Nitrate depleted beetroot juice)
- Placebo followed by Beetroot juice (Other): Placebo (70 mL nitrate depleted beetroot juice) for 14 days followed by Nitrate rich Beetroot juice for 14 days
  Interventions: Dietary Supplement: Placebo (70 mL Nitrate depleted beetroot juice) followed by 70mL Nitrate Rich Beetroot Juice

INTERVENTIONS:
Dietary Supplement: 70mL Nitrate Rich Beetroot Juice followed by placebo (Nitrate depleted beetroot juice) — 70mL Nitrate Rich Beetroot Juice for 14 days followed by placebo (Nitrate depleted beetroot juice) for 14 days
  Arms: Beetroot juice followed by placebo
Dietary Supplement: Placebo (70 mL Nitrate depleted beetroot juice) followed by 70mL Nitrate Rich Beetroot Juice — Placebo (70 mL Nitrate depleted beetroot juice) for 14 days followed by 70mL Nitrate Rich Beetroot Juice for 14 days
  Arms: Placebo followed by Beetroot juice

SUMMARY:
The purpose of this study is to see if inorganic nitrate in the form of beetroot juice helps blood flow and physical fitness in women with ANOCA and CMD. The main questions it aims to answer are:

AIM 1: Test the hypothesis that fourteen days of nitrate rich beetroot juice will increase cardiac perfusion and improve quality of life compared to placebo.

AIM 2: Test the hypothesis that fourteen days of nitrate rich beetroot juice will increase physical fitness and reduce angina and dyspnea symptoms compared to placebo.

Exploratory AIM 3: Test the hypothesis that fourteen days of nitrate rich beetroot juice will improve vascular health and function.

Participants will:

* Take study beverage for 4 weeks total.
* Stress Cardiac magnetic resonance imaging and 12 lead electrocardiograms
* Complete questionnaires
* Cycling exercise test
* Non invasive vascular testing
* Blood draws

DETAILED DESCRIPTION:
Females with heart disease often present unique phenotypes but are underrepresented in clinical trials. In females with angina, 40-65% have non-obstructive coronary artery disease (ANOCA), often due to coronary microvascular dysfunction (CMD), which represents ~52% of ANOCA cases. CMD impairs myocardial perfusion (endothelial and/or non-endothelial dysfunction), often detected as reduced coronary flow reserve (CFR). CMD is underdiagnosed despite an elevated risk for major cardiac events and current treatments for it (e.g., beta-blockers, long-acting nitrates) may confer only marginal benefits.

A critical contributor to CMD is impaired nitric oxide (NO) production, essential for vascular function. Oral inorganic nitrate (NO3-) supplementation offers a promising strategy to enhance NO bioavailability through its conversion to nitrite (NO2-) by bacteria in the mouth. NO2- acts as a precursor to NO, releasing it under hypoxic or acidic conditions commonly seen in CMD. This non-enzymatic pathway bypasses the limitations of traditional nitrate therapies, such as systemic hypotension and nitrate tolerance. Moreover, despite established benefits of physical activity ~60% of ANOCA patients experience exercise-induced angina, reduced exercise tolerance, and diminished quality of life (QoL). Recent evidence suggests, however, that exercise can increase endothelial function, endogenous NO production, LVEF, and VO2peak in ANOCA patients. Thus, increased plasma NO2- via inorganic nitrate supplementation may enhance NO delivery, promote physical activity, improve fitness and QoL in this population, which in turn may increase vascular endothelial health.

In the WISE study, >50% of women with angina had minimal or no obstructive CAD (ANOCA), yet experience worse outcomes than asymptomatic women. ANOCA involves diverse mechanisms, including coronary microvascular dysfunction (CMD), endothelial dysfunction, and vasospasm. These heterogeneities hinder responses to traditional treatments, with CMD being the most common and often linked to endothelial dysfunction.

Nitric oxide (NO) is crucial for coronary microvascular function, regulating vasodilation. In CMD, reduced NO bioavailability and endothelial nitric oxide synthase (eNOS) uncoupling impairs vasodilation and increases oxidative stress. Inflammation in CMD further exacerbates microvascular dysfunction.

Our group and others have utilized inorganic nitrate (NO3-) supplementation to increase NO bioavailability in conditions with vascular dysfunction. NO3- decreases blood pressure, arterial stiffness, oxidative stress and inflammation, while improving vascular and cardiac function. NO3- is reduced to NO under slight hypoxic or acidic conditions, common in CMD, bypassing the limitations of long-acting nitrates. ANOCA patients, a population with the high levels of initial dysfunction, may gain the most benefit from exogenous NO3-.

Dr. Allen's lab has shown that acute NO3- supplementation increases NO metabolites and augments post-exercise vascular function. Our preliminary data in postmenopausal females (PMF) also suggest a link between NO3- supplementation and reduced ET-1 and IL-6 levels compared to PL. Supplementation with NO3- may increase the "delivery pool" of NO and improve ET-1 and Il-6 dysregulation, thus augmenting vascular function, leading to improved physical function and quality of life in females with CMD.

Approach:

This will be a single-site, double-blind, randomized crossover pilot study to investigate the effects of twice daily 70 mL of beetroot juice (BTR) (~13 mmol total NO3-/day) versus PL (NO3- -depleted) in eight females. Participants with clinically stable CMD (diagnosis <2 by CMR) will be enrolled. Participants will have angina or equivalent symptoms, and no evidence of obstructive epicardial CAD (stenosis <50%) by invasive catheterization or coronary computer tomography angiography (CCTA) or FFR/CT-FFR > 0.8 within the previous 2 years.

STUDY PROCEDURES:

Participants will undergo eligibility screening and informed consent by the study coordinators. Following baseline testing, subjects will be randomized to receive consume either ∼13 mmol of NO3- (BTR) or NO3- depleted placebo (PL) daily via two (morning and night) 70-mL bottles of juice (Beet It, James White Drinks Ltd., Ipswich, UK) for 14 days. Following a 7 day washout period, participants will consume the alternate treatment (BTR or PL) for an additional 14 days.

Baseline and testing at the end of each treatment allocation will include resting vitals, fasting venous blood draw (for plasma NO3-, NO2-, ET-1, IL-6), vascular function (brachial artery flow-mediated dilation, pulse wave velocity and reflection), exercise economy testing at 2 submaximal cycle workloads, QofL questionnaires (EQ-5D-3L, Duke Activity Status Inventory, Modified Morisky Medicine Scale, Rose Dyspnea Score, and Seattle Angina Q), and stress cardiac MRI (to evaluate myocardial perfusion using dynamic first-pass imaging).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Female sex.
* Willing and able to provide written informed consent.
* Signs and symptoms of suspected ischemia prompted referral for further evaluation by cardiac catheterization or CCTA within two years of consent.
* No evidence of obstructive epicardial CAD (stenosis >50%) of a major epicardial vessel or an FFR ≤0.80 by invasive catheterization or CCTA. Patients who have not undergone cardiac catheterization of CT angiogram within the last 2 years for chest pain can be scheduled for a screening CT angiogram of the coronary arteries to confirm eligibility.
* Impaired coronary flow reserve (cut-off values depending on methodology use between ≤2.0 and ≤2.5 by stress testing PET/CMR or Invasive assessment) or Abnormal index of coronary microcirculatory resistance (e.g., IMR > 25)
* SGLT2i Naïve

Exclusion Criteria:

* History of non-ischemic cardiomyopathy LVEF <40% or hypertrophic cardiomyopathy.
* History of congestive heart failure, severe pulmonary disease, liver disease
* History of acute coronary syndrome (ACS) within previous 30 days
* Stroke within the last 180 days or intracranial hemorrhage at any time.
* Severe valvular disease
* Life expectancy <3 years, due to non-cardiovascular comorbidity.
* Pregnancy or women who are breast-feeding
* Type 1 diabetes mellitus
* Symptomatic hypotension or systolic BP<95 mmHg on 2 consecutive measurements
* Active malignancy requiring treatment at the time of visit
* Severe (eGFR <30 mL/min/1.73 m2 by CKD-EPI), unstable, or rapidly progressing renal disease at the time of randomization
* History of recurrent UTI/bladder/kidney infections
* Asthma with ongoing wheezing
* Known or suspected bronchoconstrictive or bronchospastic lung disease (ARDS, emphysema)
* Greater than first degree heart block
* Implanted cardiac device
* Profound sinus bradycardia (heart rates<40 beats per minute)
* Atrial fibrillation or supraventricular arrhythmias at time of imaging
* Known intolerance of nitrates (other than hypotension)
* History of reaction to iodinated contrast agents
* Any orthopedic, neurological, or other condition that prevents participant from exercising
* Individuals currently taking nitroglycerine (or inorganic nitrates), PDE-5 inhibitors (ex: Cialis, Viagra), and xanthine oxidase inhibitors (ex: Allopurinol)
* Smokers within the last 5 years
* Prisoners
* Cognitively impaired individuals
* Non-English Speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Coronary Flow Reserve | From enrollment to day 14
  Coronary flow reserve is calculated as the ratio of hyperemic myocardial blood flow to the resting myocardial blood flow using cardiovascular magnetic resonance myocardial perfusion imaging

SECONDARY OUTCOMES:
Submaximal Exercise Economy | From enrollment to day 14
  Submaximal Exercise Economy is calculated by a change in oxygen consumption (VO2 in mL/kg/min) from baseline to day 14.
Angina | From enrollment to day 14
  Angina is measured using the Seattle Angina Questionnaire from baseline to day 14. Question measurements range from activities being extremely limited to not at all limited by symptoms (chest pain, chest tightness, or angina) with less symptoms associated with better health related quality of life.
Dyspnea Symptoms | From enrollment to day 14
  Dyspnea symptoms are measured using the Rose Dyspnea Score comparing from baseline to day 14. Less dyspnea symptoms are associated with a better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Rodriguez-Lozano, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Hogwood AC, Ortiz de Zevallos J, Weeldreyer N, Clark JR, Mazzella V, Cain L, Myaing D, Love KM, Weltman A, Allen JD. The acute effects of exercise intensity and inorganic nitrate supplementation on vascular health in females after menopause. J Appl Physiol (1985). 2023 Nov 1;135(5):1070-1081. doi: 10.1152/japplphysiol.00559.2023. Epub 2023 Oct 5. PMID 37795531
- [Background] Hogwood AC, Ortiz de Zevallos J, Kruse K, De Guzman J, Buckley M, Weltman A, Allen JD. The effects of inorganic nitrate supplementation on exercise economy and endurance capacity across the menstrual cycle. J Appl Physiol (1985). 2023 Nov 1;135(5):1167-1175. doi: 10.1152/japplphysiol.00221.2023. Epub 2023 Sep 21. PMID 37732374
- [Background] Parker JD, Parker JO. Nitrate therapy for stable angina pectoris. N Engl J Med. 1998 Feb 19;338(8):520-31. doi: 10.1056/NEJM199802193380807. No abstract available. PMID 9468470
- [Background] Lyerly GW, Sui X, Church TS, Lavie CJ, Hand GA, Blair SN. Maximal exercise electrocardiographic responses and coronary heart disease mortality among men with metabolic syndrome. Mayo Clin Proc. 2010 Mar;85(3):239-46. doi: 10.4065/mcp.2009.0509. Epub 2010 Feb 16. PMID 20160139
- [Background] Lara J, Ashor AW, Oggioni C, Ahluwalia A, Mathers JC, Siervo M. Effects of inorganic nitrate and beetroot supplementation on endothelial function: a systematic review and meta-analysis. Eur J Nutr. 2016 Mar;55(2):451-459. doi: 10.1007/s00394-015-0872-7. Epub 2015 Mar 13. PMID 25764393
- [Background] Fejes R, Pilat N, Lutnik M, Weisshaar S, Weijler AM, Kruger K, Draxler A, Bragagna L, Peake JM, Woodman RJ, Croft KD, Bondonno CP, Hodgson JM, Wagner KH, Wolzt M, Neubauer O. Effects of increased nitrate intake from beetroot juice on blood markers of oxidative stress and inflammation in older adults with hypertension. Free Radic Biol Med. 2024 Sep;222:519-530. doi: 10.1016/j.freeradbiomed.2024.07.004. Epub 2024 Jul 5. PMID 38972612
- [Background] Kapil V, Milsom AB, Okorie M, Maleki-Toyserkani S, Akram F, Rehman F, Arghandawi S, Pearl V, Benjamin N, Loukogeorgakis S, Macallister R, Hobbs AJ, Webb AJ, Ahluwalia A. Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO. Hypertension. 2010 Aug;56(2):274-81. doi: 10.1161/HYPERTENSIONAHA.110.153536. Epub 2010 Jun 28. PMID 20585108
- [Background] Kapil V, Weitzberg E, Lundberg JO, Ahluwalia A. Clinical evidence demonstrating the utility of inorganic nitrate in cardiovascular health. Nitric Oxide. 2014 Apr 30;38:45-57. doi: 10.1016/j.niox.2014.03.162. Epub 2014 Mar 18. PMID 24650698
- [Background] Del Buono MG, Montone RA, Camilli M, Carbone S, Narula J, Lavie CJ, Niccoli G, Crea F. Coronary Microvascular Dysfunction Across the Spectrum of Cardiovascular Diseases: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 28;78(13):1352-1371. doi: 10.1016/j.jacc.2021.07.042. PMID 34556322
- [Background] Zhang Z, Li X, He J, Wang S, Wang J, Liu J, Wang Y. Molecular mechanisms of endothelial dysfunction in coronary microcirculation dysfunction. J Thromb Thrombolysis. 2023 Oct;56(3):388-397. doi: 10.1007/s11239-023-02862-2. Epub 2023 Jul 19. PMID 37466848
- [Background] Barsky L, Merz CNB, Wei J, Shufelt C, Handberg E, Pepine C, Rutledge T, Reis S, Doyle M, Rogers W, Shaw L, Sopko G. Even "WISE-R?"-an Update on the NHLBI-Sponsored Women's Ischemia Syndrome Evaluation. Curr Atheroscler Rep. 2020 Jun 18;22(8):35. doi: 10.1007/s11883-020-00852-w. PMID 32556630
- [Background] Hosadurg N, Watts K, Wang S, Wingerter KE, Taylor AM, Villines TC, Patel AR, Bourque JM, Lindner JR, Kramer CM, Sharma G, Rodriguez Lozano PF. Emerging Pathway to a Precision Medicine Approach for Angina With Nonobstructive Coronary Arteries in Women. JACC Adv. 2024 Jul 4;3(8):101074. doi: 10.1016/j.jacadv.2024.101074. eCollection 2024 Aug. PMID 39055270
- [Background] Wu Y, Zhu H, Xu Q, Li Y, Tang L. Effect of exercise training in patients with angina with nonobstructive coronary arteries: a systematic review and meta-analysis. Coron Artery Dis. 2025 May 1;36(3):252-262. doi: 10.1097/MCA.0000000000001440. Epub 2024 Oct 24. PMID 39470145
- [Background] Gulati M, Khan N, George M, Berry C, Chieffo A, Camici PG, Crea F, Kaski JC, Marzilli M, Merz CNB. Ischemia with no obstructive coronary artery disease (INOCA): A patient self-report quality of life survey from INOCA international. Int J Cardiol. 2023 Jan 15;371:28-39. doi: 10.1016/j.ijcard.2022.09.047. Epub 2022 Sep 23. PMID 36162521
- [Background] Meeder JG, Hartzema-Meijer MJ, Jansen TPJ, Konst RE, Damman P, Elias-Smale SE. Outpatient Management of Patients With Angina With No Obstructive Coronary Arteries: How to Come to a Proper Diagnosis and Therapy. Front Cardiovasc Med. 2021 Nov 2;8:716319. doi: 10.3389/fcvm.2021.716319. eCollection 2021. PMID 34796207
- [Background] Samuels BA, Shah SM, Widmer RJ, Kobayashi Y, Miner SES, Taqueti VR, Jeremias A, Albadri A, Blair JA, Kearney KE, Wei J, Park K, Barseghian El-Farra A, Holoshitz N, Janaszek KB, Kesarwani M, Lerman A, Prasad M, Quesada O, Reynolds HR, Savage MP, Smilowitz NR, Sutton NR, Sweeny JM, Toleva O, Henry TD, Moses JW, Fearon WF, Tremmel JA; Microvascular Network (MVN). Comprehensive Management of ANOCA, Part 1-Definition, Patient Population, and Diagnosis: JACC State-of-the-Art Review. J Am Coll Cardiol. 2023 Sep 19;82(12):1245-1263. doi: 10.1016/j.jacc.2023.06.043. PMID 37704315
- [Background] Wahid A, Manek N, Nichols M, Kelly P, Foster C, Webster P, Kaur A, Friedemann Smith C, Wilkins E, Rayner M, Roberts N, Scarborough P. Quantifying the Association Between Physical Activity and Cardiovascular Disease and Diabetes: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Sep 14;5(9):e002495. doi: 10.1161/JAHA.115.002495. PMID 27628572
- [Background] Banach M, Lewek J, Surma S, Penson PE, Sahebkar A, Martin SS, Bajraktari G, Henein MY, Reiner Z, Bielecka-Dabrowa A, Bytyci I. The association between daily step count and all-cause and cardiovascular mortality: a meta-analysis. Eur J Prev Cardiol. 2023 Dec 21;30(18):1975-1985. doi: 10.1093/eurjpc/zwad229. PMID 37555441
- [Background] Pinder AG, Pittaway E, Morris K, James PE. Nitrite directly vasodilates hypoxic vasculature via nitric oxide-dependent and -independent pathways. Br J Pharmacol. 2009 Aug;157(8):1523-30. doi: 10.1111/j.1476-5381.2009.00340.x. Epub 2009 Jul 7. PMID 19594749
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Jia L, Bonaventura C, Bonaventura J, Stamler JS. S-nitrosohaemoglobin: a dynamic activity of blood involved in vascular control. Nature. 1996 Mar 21;380(6571):221-6. doi: 10.1038/380221a0. PMID 8637569
- [Background] Cannon RO 3rd, Schechter AN, Panza JA, Ognibene FP, Pease-Fye ME, Waclawiw MA, Shelhamer JH, Gladwin MT. Effects of inhaled nitric oxide on regional blood flow are consistent with intravascular nitric oxide delivery. J Clin Invest. 2001 Jul;108(2):279-87. doi: 10.1172/JCI12761. PMID 11457881
- [Background] Boerhout CKM, Beijk MAM, Damman P, Piek JJ, van de Hoef TP. Practical Approach for Angina and Non-Obstructive Coronary Arteries: A State-of-the-Art Review. Korean Circ J. 2023 Aug;53(8):519-534. doi: 10.4070/kcj.2023.0109. Epub 2023 Jun 19. PMID 37525496
- [Background] Smilowitz NR, Prasad M, Widmer RJ, Toleva O, Quesada O, Sutton NR, Lerman A, Reynolds HR, Kesarwani M, Savage MP, Sweeny JM, Janaszek KB, Barseghian El-Farra A, Holoshitz N, Park K, Albadri A, Blair JA, Jeremias A, Kearney KE, Kobayashi Y, Miner SES, Samuels BA, Shah SM, Taqueti VR, Wei J, Fearon WF, Moses JW, Henry TD, Tremmel JA; Microvascular Network (MVN). Comprehensive Management of ANOCA, Part 2-Program Development, Treatment, and Research Initiatives: JACC State-of-the-Art Review. J Am Coll Cardiol. 2023 Sep 19;82(12):1264-1279. doi: 10.1016/j.jacc.2023.06.044. PMID 37704316
- [Background] Merz CN, Kelsey SF, Pepine CJ, Reichek N, Reis SE, Rogers WJ, Sharaf BL, Sopko G. The Women's Ischemia Syndrome Evaluation (WISE) study: protocol design, methodology and feasibility report. J Am Coll Cardiol. 1999 May;33(6):1453-61. doi: 10.1016/s0735-1097(99)00082-0. PMID 10334408
- [Background] Ashokprabhu ND, Quesada O, Alvarez YR, Henry TD. INOCA/ANOCA: Mechanisms and novel treatments. Am Heart J Plus. 2023 Jun;30:100302. doi: 10.1016/j.ahjo.2023.100302. Epub 2023 May 12. PMID 37377840
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Scott PE, Unger EF, Jenkins MR, Southworth MR, McDowell TY, Geller RJ, Elahi M, Temple RJ, Woodcock J. Participation of Women in Clinical Trials Supporting FDA Approval of Cardiovascular Drugs. J Am Coll Cardiol. 2018 May 8;71(18):1960-1969. doi: 10.1016/j.jacc.2018.02.070. PMID 29724348